CLINICAL TRIAL: NCT03052582
Title: Whole Milk Compared With Skimmed Milk and Effect on Lipids - A Randomized, Controlled Cross-over Study
Brief Title: Whole Milk Compared With Skimmed Milk and Effect on Lipids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: M227
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Last update posted 2018-04-02 (Actual); Status verified 2018-03

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Team 1: skimmed/whole (Active Comparator): Milktype: 3 weeks with skimmed milk followed by 3 weeks with whole milk
  Interventions: Other: Milk type
- Team 2: whole/skimmed (Active Comparator): Milktype: 3 weeks with whole milk followed by 3 weeks with skimmed milk
  Interventions: Other: Milk type

INTERVENTIONS:
Other: Milk type

SUMMARY:
The aim of the project is to investigate the effects in humans of a daily intake of whole milk compared to skimmed milk primarily and secondarily respectively on:

* Blood lipids: total-, LDL-, and HDL-cholesterol and triglycerides
* Risk markers of diabetes type 2: plasma glucose and insulin

DETAILED DESCRIPTION:
This study will be a randomized controlled 2 x 3 weeks crossover intervention study with no wash-out period, as the lipids in the blood are known to adjust after 2 weeks. The effects of a diet containing 0.5 L of whole milk (17.5 g of milk fat/day) will be compared with a diet containing 0.5 L of skimmed milk (1.5 g of milk fat/day). Blinding is not possible since the appearance of the test foods cannot be concealed. The study subjects will receive the two test foods in random order, decided by draw of lots. Blood samples will be drawn on the first day of the period and in the end of the period for each 3 week-periods.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must give their informed consent in writing, after having received oral and written information about the study

  * Age: 20-70 y
  * BMI: 18.5 - 30 kg/m2
  * Healthy men and women (with no known diseases)

Exclusion Criteria:

* Current or previous cardiovascular disease, high blood pressure or cholesterol
* Diabetes Mellitus or other severe chronic disease, including severe allergies
* Lactose intolerant or milk allergy
* Use of dietary supplements two month prior to and during the intervention Blood donations 1 month prior to and during the intervention
* Known or suspected abuse of alcohol, drugs or medication
* Pregnant or are planning pregnancy during the study period
* Extreme physical activity level (more than 10 hours tough physical activity pr. week)
* Participation in other research studies
* Inability, physically or mentally, to comply with the procedures required by the study protocol, as evaluated by the study staff

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fasting blood lipids | 3 weeks
  total, LDL and HDL cholesterol and TAG

SECONDARY OUTCOMES:
fasting plasma glucose | 3 weeks
fasting serum insulin | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tine Tholstrup, Ass Prof., Principal Investigator — Department of Nutrition, Exercise and Sports, Univeristy of Copenhagen
Locations (1):
- Department of Nutrition, Exercise and Sports, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Hansen NM, Berg P, Rix M, Pareek M, Leipziger J, Kamper AL, Astrup A, Vaarby Sorensen M, Salomo L. The New Nordic Renal Diet Induces a Pronounced Reduction of Urine Acid Excretion and Uremic Toxins in Chronic Kidney Disease Patients (Stage 3 and 4). J Ren Nutr. 2023 May;33(3):412-419. doi: 10.1053/j.jrn.2022.09.010. Epub 2022 Oct 3. PMID 36195272
- [Derived] Engel S, Elhauge M, Tholstrup T. Effect of whole milk compared with skimmed milk on fasting blood lipids in healthy adults: a 3-week randomized crossover study. Eur J Clin Nutr. 2018 Feb;72(2):249-254. doi: 10.1038/s41430-017-0042-5. Epub 2017 Dec 11. PMID 29229955